CLINICAL TRIAL: NCT07191327
Title: Testing Personalized High Definition Transcranial Direct Current Stimulation (HD-tDCS) as a Treatment of Posterior Cortical Atrophy
Brief Title: Testing Personalized High-Definition Transcranial Direct Current Stimulation (HD-tDCS) as a Treatment of Posterior Cortical Atrophy
Acronym: PCA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Benjamin Hampstead, PhD, Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUM00268033
Record Dates: First submitted 2025-09-17; First posted 2025-09-24 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Posterior Cortical Atrophy
Keywords: HD-tDCS; Functional Magnetic resonance imaging (fMRI); Positron emission tomography/computerized tomography; Memory and thinking testing; Computerized tests; Questionnaires; Blood draws; Eye tracking and vision tests; Functional Near Infrared Spectroscopy

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive sham (fake) or real stimulation for the first 4 days of HD-tDCS After the first 4 days, if participants choose to continue to be in the study, all participants will receive "real" stimulation for up to 26 weeks.
Who Masked: Participant, Investigator
Masking Description: Randomized first 4 days of treatment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Real stimulation - Randomized (Experimental): Four consecutive days (2 sessions for 20 minutes each day for a total of 8 sessions) of this blinded stimulation.
  Interventions: Device: HD-tDCS sessions
- Sham stimulation - Randomized (Sham Comparator): Four consecutive days (2 sessions for 20 minutes each day for a total of 8 sessions) of this blinded stimulation.
  Interventions: Device: Sham HD-tDCS sessions
- Real stimulation - post randomized treatment (Experimental): Participants that agree to this will have up to 26 weeks of additional HD-tDCS sessions at home or in-person.
  Interventions: Device: HD-tDCS sessions - Open-label (after randomized treatment)

INTERVENTIONS:
Device: HD-tDCS sessions — This project translates decades of observational neuroimaging research into a biologically plausible stimulation target (i.e., DAN) and uses functional magnetic resonance imaging (fMRI) and positron emission tomography (PET) to plan personalized brain stimulation and to ensure target engagement. When available; those not MRI compatible will receive a standard montage with per channel amplitudes of up to 5 milliamperes (mA) or a montage derived from other imaging methods. Participants will receive 4 days of HD-tDCS sessions in person. During these sessions participants will have electrodes placed on different areas of the head and held in place with headgear. Participants may also have memory and thinking tests during and after the sessions as well as questionnaires about the experience. Additionally, on the fourth day participants may have repeat immersive virtual reality (iVR) as well as other study activities.
  Arms: Real stimulation - Randomized
Device: Sham HD-tDCS sessions — Participants will receive 4 days of sham HD-tDCS sessions in person. During these sessions participants will have electrodes placed on different areas of the head and held in place with headgear. Participants may also have memory and thinking tests during and after the sessions as well as questionnaires about the experience. Additionally, on the fourth day participants may have repeat immersive virtual reality (iVR) as well as other study activities.
  Arms: Sham stimulation - Randomized
Device: HD-tDCS sessions - Open-label (after randomized treatment) — Optional 26 weeks of additional HD-tDCS sessions. Participants can complete up to 5 days per week, but most people will complete about 3 days per week. The study team may also collect audio recordings of these sessions. Participants can complete this in person or at-home via using a secure, HIPAA-compliant videoconferencing with the supervision of a research staff member. Participant's that decide to complete the additional sessions at home, a research staff member will train a study partner during the first 4 HD-tDCS sessions in the office. This option may not be available or appropriate for all participants and the study team member will discuss this with participant's and study partners.
  Arms: Real stimulation - post randomized treatment

SUMMARY:
This study is being completed to learn if high-definition transcranial direct current stimulation (HD-tDCS) has an effect on visual and thinking abilities in persons with posterior cortical atrophy (PCA). Participants will be randomized to receive real or sham HD-tDCS (8 sessions over 4 days).

Following the randomized treatment, participants will have optional open-label phase with real HD-tDCS up to 26 weeks and other possible testing.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis or symptoms consistent with PCA
* Fluent in English
* HD-tDCS compatible
* Stable on relevant medications for at least approximately 4 weeks prior to study enrollment
* If completing any additional, optional, long-term study visits in a remote location (i.e., not our office), a study partner is required in order to administer HD-tDCS. Those choosing to return to our office may have, but are not required to have, a study partner.

Exclusion Criteria:

* Other relevant neurological disease (e.g., epilepsy) or injuries (e.g., large vessel stroke, moderate-severe traumatic brain injury) viewed as primary to deficits since these could interfere with etiologic considerations and confound study results
* Active, relevant psychiatric conditions (e.g., bipolar disorder, schizophrenia) since the symptoms of these conditions may confound study participation.
* A recent (e.g., within the past 2 years) significant history of, or current, alcohol or drug abuse/dependence. Remote history of abuse/dependence is not exclusionary as long as it is not considered to be the primary etiology for visuospatial deficits.
* Women that are lactating/breastfeeding, pregnant, or may potentially be pregnant will be excluded from the study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2029-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Change in network connectivity measured via fMRI | Baseline and Day 5 (after 4 days of HD-tDCS)
  Functional connectivity measures whether activity in different brain regions show similar patterns of change over time. Graph theory metrics of resting-state fMRI can characterize functional connectivity within the Dorsal Attention Network (DAN).
Measure of form coherence | Baseline and at end of study intervention (up to 6 months)
  This will evaluate dorsal and ventral visual stream functioning using a visual paradigm.
Long-term change in network connectivity via fMRI | Baseline and end of study intervention (up to 6 months)
  Functional connectivity measures whether activity in different brain regions show similar patterns of change over time. Graph theory metrics of resting-state fMRI can characterize functional connectivity within the Dorsal Attention Network.
Measures of motion tasks | Baseline and at end of study intervention (up to 6 months)
  This will evaluate dorsal and ventral visual stream function. Motion coherence is measured using a visual paradigm.

SECONDARY OUTCOMES:
Measures of motion tasks | Baseline and day 5 (after 4 days of HD-tDCS)
  This will evaluate dorsal and ventral visual stream function. Motion coherence is measured using a visual paradigm.
Measure of form coherence tasks | Baseline and day 5 (after 4 days of HD-tDCS)
  Form coherence is measured using a visual paradigm.
Eye tracking - Number of fixations | Baseline and at end of study intervention (up to 6 months)
  The study team will quantify the number and duration of fixations, while the participants perform visual search, reading, or other visual tasks affected by PCA.
Eye tracking - Number of fixations | Baseline and day 5 (after 4 days of HD-tDCS)
  The study team will quantify the number and duration of fixations, while the participants perform visual search, reading, or other visual tasks affected by PCA.
Self-ratings of cognitive change using the Posterior Cortical Atrophy Questionnaire (PCA-Q) | Baseline and day 5 (after 4 days of HD-tDCS)
  The PCA-Q has 32 items and measures cognitive difficulty in 12 domains. It is reported as a composite score, with a lower overall score demonstrating less cognitive impairment.
Self-ratings of cognitive change using the Posterior Cortical Atrophy Questionnaire (PCA-Q) | Baseline and at end of study intervention (up to 6 months)
  The PCA-Q has 32 items and measures cognitive difficulty in 12 domains. It is reported as a composite score, with a lower overall score demonstrating less cognitive impairment
Immersive virtual reality (IVR) path length | Baseline and at end of study intervention (up to 6 months)
  Quotient of participants actual path length compared to the most efficient path length.
functional near infrared spectroscopy (fNIRS) - Activation magnitude of DAN (processed) | Baseline and at end of study intervention (up to 6 months)
  Measured using standard fNIRS analysis
Partner rating of cognitive change using the PCA-Q | Baseline and day 5 (after 4 days of HD-tDCS)
  The PCA-Q has 32 items and measures cognitive difficulty in 12 domains. It is reported as a composite score, with a lower overall score demonstrating less cognitive impairment
Partner rating of cognitive change using the PCA-Q | Baseline and at end of study intervention (up to 6 months)
  The PCA-Q has 32 items and measures cognitive difficulty in 12 domains. It is reported as a composite score, with a lower overall score demonstrating less cognitive impairment

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Hamstead, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Study data and documentation will be made available to the research community free of charge through the Deep Blue Data repository.
Supporting Information: Study Protocol, ICF
Time Frame: Study data will be available for sharing at the time manuscripts are published or when the grant ends, whichever is sooner. The data will be retained in Deep Blue for at least 10 years, after which it will be reviewed for continued preservation by the University Library personnel.
URL: https://deepblue.lib.umich.edu/data